CLINICAL TRIAL: NCT04676100
Title: International Cardiac Rehabilitation Registry (ICRR) Protocol
Brief Title: International CR Registry
Acronym: ICRR
Status: Enrolling by invitation | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: International Council of Cardiovascular Prevention and Rehabilitation (ICCPR (Unknown); York University (Other); Qatar University (Other)
Responsible Party: Principal Investigator, Sherry Grace, Professor, Faculty of Health & Sr. Scientist, KITE University Health Network, York University
Other Study IDs: York U ethics e2020-359; 215 (Other Grant/Funding Number: Qatar University International Research Collaboration Co-Fund 2020)
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Acute Coronary Syndrome; Heart Failure; Coronary Artery Disease
Keywords: registry; cardiac rehabilitation; mortality; equity; quality of care; patient engagement; audit and feedback; health behavior; patient-reported outcomes; depression
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure; Coronary Artery Disease; Patient Participation; Health Behavior; Depression | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiac rehabilitation — A CR program is defined as one that offers initial assessment, structured exercise (can be supervised or unsupervised) and at least one other strategy to control risk factors. The registry pertains to phase II CR.
  Quality of care and patient outcomes are benchmarked with other countries anonymously, through 2 registry dashboards (real-time). The dashboards will also show change over time in 6-month increments; Sites will be encouraged to continue to provide data on new patients until all indicators show quality as possible.
  Sites will be supported in quality improvement by the ICRR user sub-committee. High-performing programs will be recognized on ICRR's website and ICCPR's social media accounts. This mechanism may be used in future to support program accreditation.
  Other Names: quality improvement initiatives; feedback

SUMMARY:
The ICRR is a health services registry to establish the quality of CR delivery, and the effectiveness in terms of patient outcomes, in low-resource settings. The purposes of the registry are care optimization, evidentiary support for CR advocacy / policy, and research.

All programs in low-resource settings will be welcome to participate at no cost. Programs will follow procedures approved by their local ethics board for collection of program and patient-reported variables. Assessments occur pre-cardiac rehabilitation (CR), post-CR and annually thereafter.

DETAILED DESCRIPTION:
The user sub-committee has a formal site on-boarding process. Participating sites will be encouraged to enter data on all patients meeting inclusion / exclusion criteria to reduce bias. Prospective / concurrent data collection will be encouraged, to support quality improvement activities.

The company Dendrite will host the registry and ensure data security. Privacy protections will be in place, and no identifying information such as names will be entered into the registry. Data entered from sites into the registry is secured through encryption added to secure HTTP, done using Transport Layer Security. Stored data is also encrypted using InterSystems Cache database software.

There is an ICRR program survey assessing structural CR indicators. The registry variable list for patient-level data was developed based on recommendations of the Core Outcome Set-STAndards for Development (COS-STAD), through a delphi process. The final variable list and data dictionary can be found here: https://globalcardiacrehab.com/ICRR-Governance.

There are 10 program-reported variables and 16 patient-reported variables (some variables are assessed at multiple time points), assessed pre-program, post-program (dependent upon duration of each program) and each year from initial assessment (until patients expire or are unable to complete the assessments, which is ascertained by the program, or patient opt-out/withdrawal). Sites can arrange electronic data capture for the program-reported variables to contribute data to the registry, rather than manual electronic entry.

Descriptive statistics (i.e. means and standard deviations for continuous variables and frequencies with percentages for categorical variables) will be used to describe the quality of care (outcomes below). For testing change in patient outcomes pre to post-program, paired t-tests will also be used for continuous variables and chi-square test for categorical variables.

Univariate and multivariate approaches will be used to identify factors associated with outcomes, including the use of guideline-indicated therapies. Associations between patient characteristics and outcomes tested via logistic regression will be reported with odds ratios and 95% confidence intervals. Associations will be considered statistically significant when 2-sided α is <0.05. Appropriate statistical corrections for repeated measures will be performed. To limit the influence of confounding, multivariate adjustment will be used, including propensity weighting, or other techniques. Risk adjustment (e.g., socioeconomic status, indication, comorbidities, age) will be undertaken.

The registry has a data quality dashboard which displays by site completeness of data entry at each assessment point, to help reduce bias. The registry has in-built minimum and maximum values for continuous variables to reduce data entry errors. The data dictionary clearly defines each variable, and new sites are trained prior to start. The registry is being usability tested prior to launch, and piloted in Qatar. The research sub-committee will oversee a data quality process; Data audits may be supported by a registry database analyst / professional statistician.

Patient perspectives were considered in the development of the variable list and outcomes. A registry page for patients is in development (https://globalcardiacrehab.com/ICRR-for-Patients). Patients have a voice on ICRR's user sub-committee. Patients providing data pre and post-program may receive a lay summary of their progress. Lay summaries of annual registry reports may be shared with interested patients.

ELIGIBILITY:
Inclusion Criteria:

SITES:

* CR program (defined in intervention section)
* in low-resource setting (i.e., low or middle-income country according to World Bank, or in region within a higher-income country where there is under-development of CR related to financial resources, lack of healthcare system resources, lack of patient and provider awareness, and/or patient disadvantage [e.g., limited social resources, geographic barriers])

Exclusion Criteria:

SITES:

-program cannot enter data in English

PATIENTS:

* not capable to understand the registry information letter for cognitive or mental reasons (although they would also likely be excluded from CR).
* not proficient in the language of the local ethics-approved registry information letter /consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary heart disease patients who are indicated for CR are eligible for registry inclusion (e.g., acute coronary syndrome +/- revascularization, heart failure, stable coronary artery disease +/- valve or rhythm conditions); there are some exclusions to CR eligibility such as inability to ambulate.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2036-06-30 (Estimated); Study Completion 2041-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | assessed annually from initial assessment date until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  all-cause mortality, assessed via phone call
Morbidity | assessed annually from initial assessment date until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  CV event or procedure, emergency department visit for cardiac cause, or any cause hospitalization, and/or other new health condition assessed via self-report

SECONDARY OUTCOMES:
Cardiac Symptoms | assessed annually from initial assessment date until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  frequency of shortness of breath, dizziness, or chest pain in past month, assessed via self-report item (investigator-generated item based on https://www.ichom.org/portfolio/coronary-artery-disease/)
Functional capacity | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks)
  peak METs, which could be calculated based on exercise test (treadmill or bike), Duke Activity Status Index, or 6-minute walk test
Low-density lipoprotein | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks)
  in mmol/L or mg/dL from lab report
Body mass index | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks)
  weight and height will be combined to report BMI in kg/m^2
Blood pressure | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks)
  systolic and diastolic (mmHg), assessed manually or with a validated automated device
Work status | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks) & annually until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 yea
  return-to-work, if applicable, assessed via self-report of work status
Psychosocial well-being | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks) & annual until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  quality of life (Cantril's ladder) & depressive symptoms (PHQ-2)
Quality of life | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks) & annual until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  Cantril's ladder of life (10 rungs)
Depressive symptoms | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks) & annual until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  PHQ-2

OTHER OUTCOMES:
Physical activity | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks) & annual until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  self-report of minutes per week active to being at least slightly short of breath, assessed via self-report
Diet | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks) & annual until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  average number of fruits and vegetables per day, via self-report
Medication adherence | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks) & annual until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  frequency of taking heart pills as directed by physician in last month (5 point Likert scale from all the time to never), assessed via self-report
Tobacco use | pre and post-CR program (dependent upon program length, but globally the median is 8 weeks) & annual until patient expiry or withdrawal; there is no planned end date to registry but we estimate this will be assessed at 5 years
  self-report of never, current (last month), or former (use of tobacco more than 1 month prior)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry L Grace, Principal Investigator — York University & University Health Network; Karam Turk-Adawi, PhD, Principal Investigator — Qatar University
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
The ICCR will explore potential public posting of anonymous registry data in a repository in future, to augment utility of the data through availability to the scientific community.
  Specific sites may also apply for ethics approval for administrative data linkage (e.g., clinical databases, imaging or lab data, government databases or surveys), which could enable cost-effectiveness analysis for example. Contributing sites may also apply for ethics approval to survey patients over and above registry assessments.
  Any secondary use of the data for research purposes will go through separate ethical review. Requests will be vetted by the ICRR research sub-committee. No data will be released that could identify patients. This may include sharing of aggregate data on common variables with other CR registries. This research may be published in peer-reviewed journals and presented at scholarly conferences.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: to be announced
Access Criteria: The research sub-committee will develop a policy. Once approved, it will be posted at the website below
URL: https://globalcardiacrehab.com/International-CR-Registry-(ICRR)

REFERENCES:
- [Background] Poffley A, Thomas E, Grace SL, Neubeck L, Gallagher R, Niebauer J, O'Neil A. A systematic review of cardiac rehabilitation registries. Eur J Prev Cardiol. 2017 Oct;24(15):1596-1609. doi: 10.1177/2047487317724576. Epub 2017 Aug 1. PMID 28762761
- [Background] Gliklich RE, Dreyer NA, Leavy MB, editors. Registries for Evaluating Patient Outcomes: A User's Guide [Internet]. 3rd edition. Rockville (MD): Agency for Healthcare Research and Quality (US); 2014 Apr. Report No.: 13(14)-EHC111. Available from http://www.ncbi.nlm.nih.gov/books/NBK208616/ PMID 24945055
- [Background] Chowdhury MI, Turk-Adawi K, Babu AS, de Melo Ghisi GL, Seron P, Yeo TJ, Uddin J, Heine M, Saldivia MG, Kouidi E, Sadeghi M, Aljehani R, Grace SL. Development of the International Cardiac Rehabilitation Registry Including Variable Selection and Definition Process. Glob Heart. 2022 Jan 11;17(1):1. doi: 10.5334/gh.1091. eCollection 2022. PMID 35174042
- [Background] Abukhadijah HJ, Turk-Adawi KI, Dewart N, Grace SL. Qualitative study measuring the usability of the International Cardiac Rehabilitation Registry. BMJ Open. 2022 Aug 29;12(8):e064255. doi: 10.1136/bmjopen-2022-064255. PMID 36038174
- See also: Registry page for interested programs and the CR community. Patient website to be developed — https://globalcardiacrehab.com/International-CR-Registry-(ICRR)